CLINICAL TRIAL: NCT02405117
Title: A Mobile Behavioral Monitoring Intervention for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Evan Goulding, Assistant Professor, Department of Psychiatry and Behavioral Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH100460 (NIH); 1R34MH100460 (NIH)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Behavior Therapy; Technology Assisted; Mobile Phone; Smartphone
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LiveWell System (Experimental): For 16 weeks, participants will be asked to carry a mobile phone and wear a wrist-worn device for measuring activity. Participants in this arm will receive the psychosocial intervention via a smartphone and context-dependent feedback based on self-report and behavioral data. Providers whose patients are randomized to this arm will also be asked to enroll in order to receive information and notifications about patient status for the duration of the study.
  Interventions: Behavioral: LiveWell System
- Treatment As Usual (No Intervention): For 16 weeks, participants will be asked to carry a mobile phone and wear a wrist-worn device for measuring activity. Participants in this arm will be asked to provide limited self-report data via the phone.

INTERVENTIONS:
Behavioral: LiveWell System — For 16 weeks, participants will be asked to carry a mobile phone and wear a wrist-worn device for measuring activity. Participants in this arm will receive the psychosocial intervention via a smartphone and context-dependent feedback based on self-report and behavioral data. Providers whose patients are randomized to this arm will also be asked to enroll in order to receive information and notifications about patient status for the duration of the study
  Arms: LiveWell System

SUMMARY:
This study will develop and pilot a smartphone intervention, LiveWell, to enhance patient self-management of bipolar disorder and facilitate more efficient, timely care delivery by mental health providers. The intervention uses a mobile application to collect daily self-report and continuous behavioral data and adapts intervention content to create a highly tailored and user-responsive treatment system. Patient data collected by the phone will also be provided to clinicians to allow for better evaluation and targeting of treatment. The goal is to reduce symptoms and prevent relapse in patients with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a severe and chronic mental illness that significantly increases mortality and greatly impairs functioning. Despite the use of pharmacological treatments, multiple acute episodes, long episode duration, and significant inter-episode sub-syndromal symptoms are common in patients with bipolar disorder. As a result, patients with bipolar disorder are symptomatically ill about half the time. There is clear evidence that the addition of psychotherapeutic interventions to medication management improves treatment outcomes, yet only about half of bipolar patients receive combined treatment. Current therapies also have limitations in terms of: 1) reliance on subjective patient self report and 2) difficulties in identifying warning signs of impending episodes. Furthermore, direct measurement of observable daily patterns of behavior is not routinely available, even though alterations in sleep and activity are core symptoms of bipolar disorder. Improving access to and long-term engagement in psychosocial interventions is needed to substantially improve treatment.

The investigators are developing a smartphone intervention that aims to make proven psychosocial interventions for bipolar disorder more readily and routinely accessible to patients as part of their day-to-day lives. The intervention, called LiveWell, will capture and feedback data about sleep and activity to assist patients in regularizing daily rhythms as well as help them monitor, recognize, and manage early warning signs of impending mood episodes. Behavioral and self-report data collected by the phone will also be used to provide clinicians with information regarding patient clinical status. This will increase patient-provider communication and allow for better evaluation and targeting of treatment.

Participation in the study will last 4 months. All participants will first undergo initial assessments that will include a telephone interview and a face-to-face interview with a certified study psychiatrist for the purpose of confirming diagnosis. Eligible participants will then be assigned randomly to the LiveWell or TAU group. Participants assigned to either group will be provided with a smartphone and wrist-worn device, and will be asked to carry the phones with them whenever they leave home and to wear the wrist-worn devices 24-hours a day 7 days a week. Participants assigned to the LiveWell intervention will be asked to undergo a 16 week psychosocial intervention consisting of phone-based self-monitoring and educational tools to help them learn skills to better manage symptoms. Participants assigned to the TAU group will be asked to provide limited self-report data on wellness and sleep. All participants, regardless of assigned group, will be asked to participate in assessments delivered over the phone to assess presence and severity of mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Bipolar Disorder Type I.
* Minimum of 2 acute episodes in last 2 years.
* Receiving psychiatric care from a mental health provider willing to receive notifications and information regarding subject symptom status via the LiveWell system.

Exclusion Criteria:

* Not involved in current psychiatric care.
* Current substance use disorders or other psychiatric diagnosis or symptoms (e.g. dissociate disorder, psychotic symptoms) for which participation in this study is either inappropriate or dangerous.
* Pregnancy or plans to become pregnant.
* Visual impairments limiting mobile phone use.
* An inability to speak and read English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Percent Time Symptomatic | Participants will be followed for the duration of the 16 week trial.
  Percent time symptomatic will be assessed using ratings that measure the presence and severity of manic and depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Evan H. Goulding, MD PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided